CLINICAL TRIAL: NCT02550756
Title: An Open Label, Ascending Dose Study to Evaluate the Safety and Tolerability of CNTX-4975 in Subjects With Painful Intermetatarsal Neuroma (Morton's Neuroma)
Brief Title: Study to Evaluate the Safety and Tolerability of CNTX-4975 in Subjects With Painful Intermetatarsal Neuroma (Morton's Neuroma)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4975-MN-201
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Morton's Neuroma
MeSH Terms: conditions — Morton Neuroma | interventions — Capsaicin

ARMS (2):
- 0.2 mg of CNTX-4975 (Experimental): CNTX-4975 will be provided at a capsaicin concentration of 2.0 mg/ml and will be diluted to final concentration using sterile water and 30% PEG 300. Dose volume 1.0 mL-2.0 mL will be used at the discretion of the investigator. Capsaicin concentration will be 0.1 to 0.2 mg/ml
  Interventions: Drug: CTNX-4975
- 0.6 mg of CNTX-4975 (Experimental): CNTX-4975 will be provided at a capsaicin concentration of 2.0 mg/ml and will be diluted to final concentration using sterile water and 30% PEG 300. Dose volume 1.0 mL-2.0 mL will be used at the discretion of the investigator. Capsaicin concentration will be 0.3 to 0.6 mg/ml
  Interventions: Drug: CTNX-4975

INTERVENTIONS:
Drug: CTNX-4975
  Other Names: Capsaicin

SUMMARY:
The purpose of this study is to confirm that the local anesthetic applied to subjects with Morton's Neuroma satisfactorily mitigates procedure pain and ensures that post-procedure discomfort or pain will not result in bias or breaking of the blind in the planned Phase 2b study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged >/=18 years at the time of the Screening Visit.
2. Symptoms of intermetatarsal neuroma for at least 30 days prior to the Screening Visit.
3. Diagnosis of intermetatarsal neuroma (Morton's neuroma) based on medical history and physical examination with evidence of focal tenderness and pain in the area of the neuroma, confirmed by ultrasound or other imaging modality. Typically the subject will have sensory symptoms in the distribution of the affected common digital nerve. However, provided the imaging study is positive, the presence of these sensory symptoms is not required. The neuroma may be in either the second or third intermetatarsal space.
4. An average pain score of 4.0 to 9.0 (during the 7 days prior to dosing) on the Numeric Pain Rating Scale (NPRS), as rated daily at bedtime for average pain while walking in the last 24 hours, relevant to the affected foot. At least 4 of 7 scores during the week prior to dosing must be recorded.
5. For female subjects: reproductive status is such that the subject is surgically sterile, at least 2 years postmenopausal, or using a medically acceptable method of birth control; if of child-bearing potential, is not pregnant (negative urine pregnancy test prior to enrollment), is not planning to get pregnant during the course of the study, and is not lactating.
6. Willing and able to understand the study requirements, abide by the study restrictions, complete the study procedures, pain scales, and diaries, and to communicate meaningfully with the study personnel.
7. Signed an Informed Consent Form approved by the Institutional Review Board.

Exclusion Criteria:

1. Clinically significant bursitis or another significant symptomatic condition in the region of or adjoining the neuroma.
2. The subject has more than one intermetatarsal neuroma on the foot to be injected (index foot).
3. Prior use of injection with a sclerosing agent such as alcohol or phenol, or prior surgery for intermetatarsal neuroma on the affected foot.
4. Prior injection of corticosteroid in the index foot or oral use of corticosteroids within 30 days of screening.
5. The subject has another painful condition that, in the judgment of the investigator, would interfere with the subject's ability to evaluate the pain and functional limitations that arise from the intermetatarsal neuroma.
6. Other painful foot pathology (e.g., bunion, hammertoe, plantar fasciitis, etc.) or evidence of clinically meaningful ischemia which in the opinion of the investigator would interfere with evaluation of the symptoms and functional limitations that arise from the intermetatarsal neuroma. For example, if the subject has pain from a bunion but that pain is easily distinguished by the subject from the neuroma pain, then the subject would still be a candidate for the study. Note, however, that the subject should also be able to distinguish the neuroma pain from the bunion pain in terms of foot function. In general, if another foot pain condition (in the same foot) gives rise to pain that is greater than the neuroma pain, then that subject should in most instances be excluded.
7. Signs of arterial insufficiency in the feet.
8. Ulcer and/or wound in the foot affected by the neuroma.
9. Active cutaneous disease, or other anatomical or physiological foot disorder, at the anticipated site of study drug injection.
10. History of clearly documented allergic reaction to local anesthetics or capsaicin.
11. Presence of any medical condition or instability that, in the judgment of the Investigator, might adversely impact the conduct of the study or resulting data, including chronic conditions that are likely to alter the rate of healing or are likely to result in safety complications unrelated to the study medication, such as uncontrolled diabetes mellitus or vascular disease.
12. Clinically significant laboratory result at the Screening Visit (in the opinion of the Investigator).
13. Has diabetic neuropathy or other length dependent neuropathy.
14. Use of any investigational medication in the 30 days prior to the current study, is scheduled to receive such an agent while participating in this study, or received a topical or injected investigational medication in the index foot within the past 60 days.
15. Use of topical medication on the index foot within 7 days of screening (including lidocaine or capsaicin).
16. Prior participation in an ALGRX 4975 study.
17. History of substance abuse disorder within the past year as defined by DSM-IV, has current evidence for a substance abuse disorder, is receiving medicinal treatment for drug abuse, or tests positive upon urine drug screen for a substance of abuse.
18. Has any condition or is taking any medication that would be contraindicated for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of a single injection of CNTX-4975 through assessment of incidence, intensity, relationship and seriousness of treatment-emergent adverse events | up to 6 months post injection
Evaluate the safety and tolerability of a single injection of CNTX-4975 through treatment-emergent changes in vital signs and laboratory tests | up to 2 weeks post injection
  blood pressure, hart rate, respiration rate, body temperature, weight
Evaluate the safety and tolerability of a single injection of CNTX-4975 through treatment-emergent changes in sensory and motor examination of the foot | up to 6 months post injection
  Light touch and pin prick of toes in both feet and evaluation of flexion and extension ability
Evaluate the safety and tolerability of a single injection of CNTX-4975 through treatment-emergent changes at injection site by Injection site assessment 5-point scale for erythema and edema | 1, 2, and 4 hours post injection

SECONDARY OUTCOMES:
Evaluate the magnitude and duration of analgesic efficacy of CNTX-4975 using Numeric Pain Rating Scale (NPRS, 0-10 scale) | Up to 6 months post injection
Evaluate Patient Global Impression of Change (PGIC) | Up to 6 months post injection
Evaluate functional improvement based on Manchester Foot Pain and Disability Index (MFPDI) | 2 weeks post injection